CLINICAL TRIAL: NCT04903132
Title: Cellular Senescence and Its Contribution to COVID-19 Long-Hauler Syndrome
Brief Title: Cellular Senescence and COVID-19 Long-Hauler Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-011877
Record Dates: First submitted 2021-05-24; First posted 2021-05-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Longhauler's Syndrome Cohort: Subject's with longhaulers
- Control Cohort: Control cohort will not have had a known case of COVID-19 or Longhauler's syndrome
- COVID Control Cohort: Subjects who have had COVID-19 but no known Longhauler's syndrome

SUMMARY:
The purpose of this study is to test if senescent cells and their secretome contribute to Long-Hauler Syndrome and if a clinical trial of senolytic drugs, which selectively eliminate senescent cells, should be initiated.

ELIGIBILITY:
Longhauler's Cohort -

Inclusion Criteria:

* Ability to give informed consent or LAR.
* At least 18 years old.
* Ability of subject or LAR to read and speak the English language.
* Positive PCR or antibody test within 12 months of initial study visit.
* Patient of the Long-Hauler Syndrome clinic and differential diagnosis of Long-Hauler Syndrome.

Exclusion Criteria:

* Any potential participant who refuses medical record review.
* Pregnant females.
* Incarcerated individuals.
* Inability to cooperate or any medical condition that, in the opinion of the investigator, interferes with the evaluation of the study objectives or increases the subject's risk by participating in the study.

Control Cohort -

Inclusion Criteria:

* Ability to give informed consent
* At least 18 years old
* Ability of subject to read and speak the English language

Exclusion Criteria:

* Known case of COVID-19.
* Any potential participant who refuses medical record review.
* Pregnant females.
* Incarcerated individuals.
* Inability to cooperate or any medical condition that interferes with the evaluation of the study objectives or increases the subject's risk by participating in the study.

COVID-19 Control Cohort

Inclusion Criteria:

* Ability to give informed consent.
* At least 18 years old.
* Ability of subject to read and speak the English language.
* Known case of COVID-19.

Exclusion Criteria:

* Known Longhauler's syndrome/Post-COVID
* Any potential participant who refuses medical record review.
* Pregnant females.
* Incarcerated individuals.
* Inability to cooperate or any medical condition that interferes with the evaluation of the study objectives or increases the subject's risk by participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Longhauler's Cohort: Patients must be at least 18 years or older, have a positive PCR or antibody test within six months, and report any ongoing symptoms associated with Post-COVID or Long-Haulers Syndrome.
  Control Cohort: Patients must be at least 18 years or older, have not had a known case of COVID-19 or Longhauler's syndrome.
  COVID Control Cohort: Patients must be at least 18 years or older and have had COVID-19 but no known Longhauler's syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between features of Long-Hauler Syndrome with markers of cellular senescence and SASP factors | 6 months
  If a correlation between features of Long-Hauler Syndrome with markers of cellular senescence and SASP factors can be demonstrated, or SASP factors are higher in Long-Hauler Syndrome clinic patients than age- and sex-matched controls (using archived samples) in this pilot study, a protocol will be submitted to the IRB for a trial in Long-Hauler Syndrome patients of senolytic drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T. Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials